CLINICAL TRIAL: NCT00865605
Title: A Single-blind, Single Exposure Study, to Evaluate the Vasoconstriction Activity of Topically Delivered Halobetasol Propionate Ointment in Normal Skin in Healthy Adult Subjects: Pivotal Bioequivalence Study
Brief Title: Pivotal Bioequivalence Study of Topically Delivered Halobetasol Propionate Ointment in Normal Skin in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Christine Winslow, Director of Clinical Development, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: DP03-689
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: bioequivalence; Vasoconstriction; Halobetasol; Healthy subjects
MeSH Terms: interventions — halobetasol; Ointments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Halobetasol Propionate 0.05% Ointment, single exposure
  Interventions: Drug: Halobetasol Propionate 0.05% Ointment, single exposure
- B (Active Comparator): Ultravate® 0.05% ointment, single exposure
  Interventions: Drug: Ultravate® 0.05% ointment, single exposure

INTERVENTIONS:
Drug: Halobetasol Propionate 0.05% Ointment, single exposure — A: Other Subjects received Alpharma/Purepac USHP formulated products
  Other Names: Halobetasol
  Arms: A
Drug: Ultravate® 0.05% ointment, single exposure — Subjects received Bristol-Myers Squibb Company formulated products
  Other Names: Halobetasol
  Arms: B

SUMMARY:
The purpose of this study is to compare the vasoconstriction response profile and bioequivalence between one innovator lot of Ultravate® 0.05% ointment and one test/generic lot of Halobetasol propionate 0.05% ointment (Alpharma USPD, Inc.).

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: A single blind, single-exposure study on healthy adult male and female subjects.

Official Title: A Single-blind, Single Exposure Study, to Evaluate the Vasoconstriction Activity of Topically Delivered Halobetasol Propionate Ointment in Normal Skin in Healthy Adult Subjects: Pivotal Bioequivalence Study

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Vasoconstrictor Response

ELIGIBILITY:
Inclusion Criteria:

* Subject understands the study, is willing to participate, and gives written informed consent.
* Subject demonstrates adequate vasoconstriction to the screening topical corticosteroid Halobetasol propionate 0.05% ointment within 30 days of dosing.
* Subject is a non-smoking (minimum of 14 days), male or female, ages of 18 - 65 years, inclusive.
* Subject is within 20% of their ideal body weight as defined by the 1999 Metropolitan Life Insurance Company Height and Weight Tables.
* Subject is judged by the Investigator to be healthy on the basis of pre-study medical history.
* Subjects of child-bearing potential agree to use an acceptable method of birth control during study participation (e.g. abstinence, any prescribed birth control method, double barrier method, Le. condom plus foam, condom plus diaphragm).
* Subject is willing to refrain from excessive consumption of sodium in food or beverage 48hrs before and for the duration of the study.
* Subject is willing to shower using the same soap/cleansers for the duration of the study.
* Subject is willing to follow study restrictions.

Exclusion Criteria:

* Subject has a past or current medical condition that might significantly affect pharmacodynamic response to topical corticosteroids.
* Subject has diabetes mellitus, clinically significant hypertension or circulatory disease.
* Subject is taking any medication on a regular basis that could modulate blood flow (constrictor or dilator), with the exception of any prescribed birth control method and hormone replacement therapy. Examples of such drugs include nitroglycerin, anti- hypertensives, antihistamines, NSAIDs, aspirin, phenylpropanolamine, phentolamine or any other medications deemed inappropriate by the Investigator.
* Subject is planning to use any exclusionary over-the-counter (OTC) medications within 48 hours prior to or throughout the study that could modulate vascular blood flow.
* Subject intends to start, stop or change dose of any prescription or OTC medication within 48 hours prior to or throughout the study. Acetaminophen may be administered, if needed.
* Subject has used prescription or OTC topical medications on the ventral forearms within 1 month prior to study conduct.
* Subject has a history of sensitivity/allergy to the ingredients found in the test formulations or has a history of adverse reactions to topical or systemic corticosteroids.
* Subject has a significant history of allergy to soaps, lotions, emollients, ointments, creams, cosmetics, adhesives, or latex.
* Subject has a history of significant skin conditions or disorders, for example, psoriasis, atopic dermatitis, etc.
* Subject has a history of significant dermatologic cancers, for example, melanoma or squamous cell carcinoma. Basal cell carcinomas that were superficial and do not involve the investigative site are acceptable.
* Subject has an obvious difference in skin color between arms or the presence of a skin condition, scar tissue, tattoo or coloration that would interfere with placement of test sites, their assessments, their reaction to drug or could compromise the safety of the subject.
* Subject has used topical medications on the ventral forearms within 1 month prior to dosing.
* Subject has used a tobacco product within 14 days of study conduct.
* Subject has a clinically significant history of drug abuse or alcoholism.
* Subject has donated or received blood within 30 days prior to dosing.
* Subject's caffeine intake is greater than 500 mg per day (1 cup of coffee contains approximately 85 mg of caffeine).
* Subject is unwilling to abstain from alcohol or caffeine for 48 hours prior to and throughout the study.
* (Females only): Subject is pregnant or lactating.
* Subject has participated in another investigational drug, medical device, or biologics study within 30 days prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2003-12; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Vasoconstrictor Response | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Lehman,, M.Sc., Principal Investigator — DermTech International
Locations (1):
- DermTech International, San Diego, California, United States